CLINICAL TRIAL: NCT02971007
Title: A Multi-Center Randomized Study to Evaluate the Safety, Tolerability, and Efficacy of Oral Encochleated Amphotericin B (CAMB/MAT2203) Compared With Oral Fluconazole in the Treatment of Moderate to Severe Vulvovaginal Candidiasis (VVC)
Brief Title: Safety and Efficacy of Oral Encochleated Amphotericin B (CAMB/MAT2203) in the Treatment of Vulvovaginal Candidiasis (VVC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Matinas BioPharma Nanotechnologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MB-70005
Record Dates: First submitted 2016-11-10; First posted 2016-11-22 (Estimated); Results first posted 2018-10-05 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Vulvovaginitis; Yeast Infection; Yeast Infection Vaginal; Candidiasis, Vulvovaginal
MeSH Terms: conditions — Vulvovaginitis; Candidiasis, Vulvovaginal | interventions — Fluconazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CAMB 200 mg (Experimental): 200 mg CAMB (MAT2203) Oral Amphotericin B
  Interventions: Drug: Oral Encochleated Amphotericin B (CAMB)
- CAMB 400 mg (Experimental): 400 mg CAMB (MAT2203) Oral Amphotericin B
  Interventions: Drug: Oral Encochleated Amphotericin B (CAMB)
- Fluconazole 150 mg (Active Comparator): Fluconazole Diflucan
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Oral Encochleated Amphotericin B (CAMB) — lipid-crystal nano-particle formulation amphotericin B
  Other Names: MAT2203
  Arms: CAMB 200 mg; CAMB 400 mg
Drug: Fluconazole
  Arms: Fluconazole 150 mg

SUMMARY:
This is a multi-center, randomized study to evaluate the safety, tolerability, and efficacy of 200 mg CAMB and 400 mg CAMB compared with a single 150 mg dose of fluconazole in the treatment of moderate to severe VVC.

DETAILED DESCRIPTION:
This is a multi-center, randomized study to evaluate the safety, tolerability, and efficacy of 200 mg CAMB and 400 mg CAMB compared with a single 150 mg dose of fluconazole in the treatment of moderate to severe VVC.

Approximately 75 women with moderate to severe VVC will be randomized to 1 of 3 treatment groups (200 mg CAMB, 400 mg CAMB, or fluconazole) to achieve approximately 25 subjects in each group. The primary objective of this study is to evaluate the safety of 200 mg and 400 mg doses of oral CAMB for 5 days compared with a single 150 mg dose of oral fluconazole in subjects with moderate to severe VVC. The secondary efficacy objectives of this study included the clinical cure rate, mycology eradication and responder outcome. Tertiary objectives include pharmacokinetics.

ELIGIBILITY:
Key Inclusion Criteria:

Informed consent

Clinical diagnosis of moderate to severe VVC

Negative pregnancy test

Vaginal pH less than 4.5

Key Exclusion Criteria:

Has an intolerance or hypersensitivity to any amphotericin B (AMB) product, or to azole antifungal drugs

Receiving antifungal therapy unrelated to VVC or has evidence of systemic fungal infections requiring antifungal therapy

Has received treatment for VVC within the past 30 days or has experienced 4 or more episodes of VVC in the past 12 months

Has another cause of vulvovaginitis

Has other urogenital infection(s) that would potentially alter their response to disease

Has another vaginal or vulvar condition that would confound the interpretation of clinical response

Has significant laboratory abnormality at screening

Has any known azole-resistant Candida infection;

Has any other condition the Investigator believes would interfere with the subject's ability to provide informed consent, comply with study instructions, or puts the subject at undue risk

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Kling, Study Director — Matinas BioPharma Nanotechnologies, Inc.
Locations (23):
- United States (23):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Precision Trials, LLC, Phoenix, Arizona
  - National Research Institute - Wilshire, Los Angeles, California
  - South Florida Medical Research, Aventura, Florida
  - Neostart Corporation dba AGA Clinical Trials, Hialeah, Florida
  - Altus Research, Lake Worth, Florida
  - Advanced Research Institute Inc, New Port Richey, Florida
  - Healthcare Clinical Data, Inc., North Miami, Florida
  - Clinical Research of West Florida - Tampa, Tampa, Florida
  - Visions Clinical Research, Wellington, Florida
  - Mt. Vernon Clinical Research - Wake Research, Atlanta, Georgia
  - Brighton Clinical Research Associates, Norcross, Georgia
  - Medpharmics, Metairie, Louisiana
  - New England Center for Clinical Research, Inc., Fall River, Massachusetts
  - Lawrence OB/GYN, Lawrenceville, New Jersey
  - ProHEALTH Care Associates, LLC - Suffolk OB-GYN, Port Jefferson, New York
  - PMG Research of Salisbury, LLC., Salisbury, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Complete Health Care for Women, Columbus, Ohio
  - Study Center, Columbus, Ohio
  - Jackson Clinic, Jackson, Tennessee
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Tidewater Clinical Research, Inc., Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period November 2016 to May 2017 at 22 medical clinics in USA
Pre-assignment Details: Enrolled patients were excluded from the study before assignment to groups due to abnormal laboratory test results, negative potassium hydroxide test (KOH) for vaginal yeast or vaginal pH greater than 4.5 during the screening process.
Groups:
- Fluconazole 150 mg: Fluconazole Diflucan
  Fluconazole
Period: Overall Study
Arm/Group | CAMB 200 mg | CAMB 400 mg | Fluconazole 150 mg
Started | 46 | 45 | 46
Completed | 44 | 42 | 45
Not Completed | 2 | 3 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Patient had yeast at Day 5 visit | 1 | 0 | 0
Not completed — Patient discontinued study drug | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CAMB 200 mg | CAMB 400 mg | Fluconazole 150 mg | Total
Number analyzed (Participants) | 46 | 45 | 46 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (12.63) | 36.2 (9.77) | 34.3 (11.25) | 35.4 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 45 | 46 | 137
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 14 | 9 | 43
  Not Hispanic or Latino | 26 | 31 | 37 | 94
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 22 | 24 | 58
  White | 34 | 23 | 22 | 79
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 46 | 45 | 46 | 137
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 30.49 (8.136) | 30.64 (8.411) | 29.50 (6.973) | 30.21 (7.819)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Outcome Assessed at Test of Cure Visit
Description: Number of patients determined to be a Clinical Cure (resolution of the VVC signs and symptoms that were present at baseline without further antifungal treatment); Clinical Failure (incomplete resolution of signs and symptoms of VVC that were present at baseline or new signs and symptoms have developed and require the initiation of non-study antifungal drugs); or Clinical indeterminate (insufficient data are available to determine if the subject is a cure or failure)
Time Frame: 12 days
Population: All randomized participants who had a Candida species isolated on culture of vaginal specimen at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | CAMB 200 mg | CAMB 400 mg | Fluconazole 150 mg
Number analyzed (Participants) | 25 | 22 | 32
Participants
  Clinical Cure | 13 | 12 | 24
  Clinical Failure | 12 | 8 | 7
  Clinical Indeterminate | 0 | 2 | 1
Statistical Analysis 1: Comparison: CAMB 200 mg vs CAMB 400 mg vs Fluconazole 150 mg; No formal sample size calculations were made. The sample size was determined empirically rather than with a specific statistical rationale and is considered sufficient to achieve the study objectives of this proof of concept study. Women with moderate to severe Vulvovaginal candidiasis were randomized in a 1:1:1 ratio to 1 of 3 treatment groups, stratified by signs and symptoms composite score of up to 12 (moderate) and greater than 13 (severe); Test type: Other — Statistical analyses primarily descriptive with no formal statistical hypothesis testing. Summary statistics are presented by treatment group. For continuous variables, the number of observations, mean, standard deviation, median, minimum and maximum are provided as summary statistics; Statistical analyses primarily descriptive with no formal statistical hypothesis testing. Summary statistics are presented by treatment group. For continuous variables, the number of observations, mean, standard deviation, median, minimum and maximum are provided as summary statistics

2. Secondary Outcome: Mycological Outcome Assessed at Test of Cure
Description: Number of patients with mycological eradication (vaginal swab culture negative for growth of baseline Candida species); mycological persistence (vaginal swab culture positive for growth of baseline Candida species); or mycological indeterminate (vaginal swab culture not available or the culture cannot be interpreted or is considered contaminated)
Time Frame: 12 days
Population: All randomized participants who had a Candida species isolated on culture of vaginal specimen at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | CAMB 200 mg | CAMB 400 mg | Fluconazole 150 mg
Number analyzed (Participants) | 25 | 22 | 32
Participants
  Mycological Eradication | 9 | 7 | 27
  Mycological Persistence | 16 | 13 | 4
  Mycological Indeterminate | 0 | 2 | 1

3. Secondary Outcome: Overall Response
Description: Number of patients with overall response at Day 12 (Test of cure visit) of composite signs and symptoms defined as overall success (achievement of both a clinical cure and microbiological eradication); overall failure (clinical failure or microbiological persistence) or overall indeterminate (insufficient data are available to determine if the patient is an overall success or failure).
Time Frame: 12 Days
Population: All randomized participants who had a Candida species isolated on culture of vaginal specimen at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | CAMB 200 mg | CAMB 400 mg | Fluconazole 150 mg
Number analyzed (Participants) | 25 | 22 | 32
Participants
  Overall Success | 4 | 3 | 22
  Overall Failure | 21 | 17 | 9
  Overall Indeterminate | 0 | 2 | 1

4. Secondary Outcome: Change in Composite Clinical Cure Score
Description: The percent change from baseline to Day 12 (Test of Cure Visit) of the composite clinical cure score of signs (erythema, edema or excoriation) and symptoms (itching, burning or irritation) on a scale of 0 to 3 for each sign and symptom where 0 = none (complete absence of any sign or symptom); 1 = mild (slight); 2 = moderate (definitely present) or 3 = severe (marked/intense). The maximum score at baseline = 18 (score of 3 for each sign and symptom). The minimum score at baseline = 4 (score of 2 for at least 2 signs or symptoms). A lower score at Day 12 represents a better outcome.
  The mean percent change from baseline score to Day 12 score is presented for each arm as a negative number and represents a decrease in severity of signs and symptoms. A bigger decrease represents a better outcome.
Time Frame: Between randomization visit (Baseline) and Day 12 visit (Test of Cure)
Population: All randomized participants who had a Candida species isolated on culture of vaginal specimen at baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CAMB 200 mg | CAMB 400 mg | Fluconazole 150 mg
Number analyzed (Participants) | 25 | 22 | 32
percent change | -80.9 (24.63) | -80.1 (44.66) | -94.0 (13.71)

ADVERSE EVENTS:
Time Frame: Adverse event data collected from randomization through follow-up phone call between Day 21 to Day 30.
Arm/Group | CAMB 200 mg | CAMB 400 mg | Fluconazole 150 mg
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/45 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/45 | 0/46
Other Adverse Events (participants affected / at risk) | 10/46 | 12/45 | 4/46
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAMB 200 mg (N=46) | CAMB 400 mg (N=45) | Fluconazole 150 mg (N=46)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Bacterial Vaginosis (Infections and infestations) | 3 (3) | 5 (5) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
This is a proof of concept study not designed or powered to support an indication for the treatment of VVC but to establish safety, tolerability and efficacy in a non-life threatening fungal infection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data may be considered for publication in a scientific journal or for reporting at a scientific meeting. Each Investigator is obligated to keep data pertaining to the study confidential and must consult with the Sponsor before any study data are submitted for publication. Sponsor reserves the right to deny publication rights until mutual agreement on the content, format, interpretation of data in the manuscript, and journal selected for publication are achieved.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/07/NCT02971007/Prot_SAP_000.pdf